CLINICAL TRIAL: NCT03152058
Title: Certolizumab to Prevent Pregnancy Complications in High-Risk Patients With APS or SLE - (IMPACT Study: IMProve Pregnancy in APS With Certolizumab Therapy)
Brief Title: IMPACT Study: IMProve Pregnancy in APS With Certolizumab Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David Ware Branch (Other)
Collaborators: Hospital for Special Surgery, New York (Other); University of Toronto (Other); NYU Langone Health (Other)
Responsible Party: Sponsor-Investigator, David Ware Branch, MD, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 94818
Record Dates: First submitted 2017-05-01; First posted 2017-05-12 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: High Risk Pregnancy; Pregnancy Complications; Antiphospholipid Syndrome in Pregnancy; Lupus Anticoagulant Disorder
MeSH Terms: conditions — Pregnancy Complications | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Certolizumab Pegol (Experimental): All participants are administered certolizumab [400 mg (given as two subcutaneous injections of 200mg) initially and 2 and 4 weeks later, followed by 200 mg every other week thereafter.
  1st dose of certolizumab will be administered by 8 weeks and 6 days gestation and discontinued at 27 weeks 6 days.
  The regimen of heparin and low dose aspirin is a standard of care treatment for this patient population and is not considered part of the research intervention.
  Interventions: Drug: Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab Pegol — Certolizumab [400 mg (given as two subcutaneous injections of 200mg) initially and 2 and 4 weeks later, followed by 200 mg every other week thereafter] The 1st dose of certolizumab will be administered by 8 weeks and 6 days gestation and discontinued at 27 weeks 6 days.
  The regimen of heparin and low dose aspirin is a standard of care treatment for this patient population and is not considered part of the research intervention.
  Other Names: Cimzia

SUMMARY:
This treatment trial evaluates the addition of an anti-tumor necrosis factor-alpha drug, certolizumab, to usual treatment (a heparin agent and low-dose aspirin) in pregnant women with antiphospholipid syndrome (APS) and repeatedly positive tests for lupus anticoagulant (LAC) to determine if this regimen will improve pregnancy outcomes. All enrolled patients will receive certolizumab, and pregnancy outcomes will be compared to those of women with APS and repeatedly positive tests for LAC enrolled in a previous study by the investigators.

DETAILED DESCRIPTION:
Antiphospholipid syndrome (APS) is an autoimmune disorder that occurs most commonly in women of reproductive-age and is associated with thrombosis and adverse pregnancy outcomes (APOs), such as fetal loss and preterm birth due to severe preeclampsia (PE) or placental insufficiency (PI). Traditional therapy for APS during pregnancy has been a heparin agent and low dose aspirin. However, in PROMISSE, a prospective observational study of 724 patients, 44% of pregnancies in women with APS and LAC resulted in APOs despite treatment with heparin and low dose aspirin.

The APOs in women with APS and LAC are due to failure of adequate vascularization of the developing placenta and subsequent inadequate blood flow to the placenta and fetus. Mouse models of APS show that poor placental vascularization in APS is a result of inflammation in the placenta. This inflammation leads to recruitment of neutrophils and release of more inflammatory mediators and anti-angiogenic factors. In the mouse model tumor necrosis factor-alpha is a critical downstream effector of abnormal placental development and fetal damage, and tumor necrosis factor-alpha blockade during pregnancy restores angiogenic balance, normalizes placental vascularization, and rescues pregnancies.

Based on our observations in PROMISSE and the favorable results of tumor necrosis factor-alpha blockade in our mouse models, we hypothesize that tumor necrosis factor-alpha blockade will significantly decrease the rate of fetal death and preterm delivery due to PE and PI in women with APS and LAC. The study investigators aim to determine whether tumor necrosis factor-alpha blockade during pregnancy, added to a regimen of heparin and low dose aspirin, (1) reduces the rate of APOs in women with clinical APS and LAC, and (2) alters angiogenic markers of poor placental vascularization. Investigators will conduct an open label trial of certolizumab (a tumor necrosis factor-alpha inhibitor that does not cross the placenta). The regimen of heparin and low dose aspiring is a standard of care treatment for this patient population and is not considered part of the research intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant as defined by positive test for elevated ß-HCG and having a live, appropriate sized embryo by ultrasound, but <8 weeks gestation;
* Antiphospholipid syndrome (APS);
* Positive for LAC on two or more occasions greater than 12 weeks apart within the previous 18 months. If a candidate for the study is newly diagnosed (<12 weeks) with APS, meets clinical criteria for APS and has one positive LAC confirmed by review of the medical record, she may be consented and screened. At baseline, LAC will be measured at the study core lab and she will be enrolled if it is found to be positive. The LAC measurement will be repeated 12 weeks after the initial determination and, if positive, she will remain in the study.
* Age 18-40 (+364 days) years of age and able to give informed consent
* Laboratory hematocrit >26% at time of screening.

the diagnosis of APS and LAC will be confirmed by one of the Co-PI's for each case by a review of the medical records.

Exclusion Criteria:

* Hypertension (BP >140/90) present at screening;
* Multifetal gestation;
* Type 1 or Type 2 diabetes antedating pregnancy;
* SLE patients requiring prednisone >10 mg/day;
* Platelet count <100,000 per microliter;
* Women currently taking prednisone greater than 10 mg daily for an autoimmune disorder, other than immune thrombocytopenia;

  a. More than 60 mg once daily in a tapering regimen or 20 mg once daily in a maintenance regimen for immune thrombocytopenia
* Women with urinary excretion with greater than 500 mg (0.5 g) per day (spot urine protein/creatinine ration 0.5);
* Serum creatinine >1.2 mg/dL
* History of tuberculosis or untreated positive PPD;
* Women with a tuberculin skin test induration of 5 mm or greater; or positive quantiFERON-gold test
* Women with HIV, Hepatitis B or Hepatitis C positive status;
* Known contraindications or relative contraindications to certolizumab:

  1. Active infection, e.g., chronic hepatitis B
  2. History of recurrent infection, e.g., recurrent cellulitis, or opportunistic infection
  3. History of prior active/treated endemic mycoses in the last two years (including coccidioidomycosis, blastomycosis, or histoplasmosis)
  4. History of heart failure
  5. History of peripheral demyelinating disease or Guillian-Barre syndrome
  6. History of hematologic malignancy
  7. Prior adverse reaction to certolizumab or o ther anti-TNF-α agent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility includes only pregnant women
Enrollment: 55 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fetal death and/or preterm delivery (<34 weeks) due to PE or PI in women with APS and LAC | 8 weeks gestation through 6-weeks postpartum
  Either of the following will constitute a primary outcome:
  1. Fetal death (>10 wks gestation)
  2. Severe preeclampsia or placental insufficiency requiring delivery prior to 34 weeks gestation.

SECONDARY OUTCOMES:
Additional adverse outcomes or pertinent concerns, possibly related to study intervention | 8 weeks gestation through 6-weeks postpartum
  Any one of the following is considered a secondary outcome:
  1. Neonatal death due to complications of prematurity because of preterm delivery for PE or PI
  2. Preterm labor or preterm rupture of membranes resulting in delivery prior to 36 weeks gestation
  3. PE or PI not requiring delivery prior to 34 weeks gestation
  4. Gestational age at delivery
  5. Maternal thrombosis
  6. Small-for-gestational age birthweight (<10th percentile)
  7. Known adverse reactions to certolizumab.

CONTACTS AND LOCATIONS:
Overall Officials: D. Ware Branch, MD, Principal Investigator — University of Utah
Locations (3):
- United States (2):
  - Hospital for Special Surgery, New York, New York
  - University of Utah, Salt Lake City, Utah
- TRIO Advancing Reproductive Care, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miyakis S, Lockshin MD, Atsumi T, Branch DW, Brey RL, Cervera R, Derksen RH, DE Groot PG, Koike T, Meroni PL, Reber G, Shoenfeld Y, Tincani A, Vlachoyiannopoulos PG, Krilis SA. International consensus statement on an update of the classification criteria for definite antiphospholipid syndrome (APS). J Thromb Haemost. 2006 Feb;4(2):295-306. doi: 10.1111/j.1538-7836.2006.01753.x. PMID 16420554
- [Background] Committee on Practice Bulletins-Obstetrics, American College of Obstetricians and Gynecologists. Practice Bulletin No. 132: Antiphospholipid syndrome. Obstet Gynecol. 2012 Dec;120(6):1514-21. doi: 10.1097/01.AOG.0000423816.39542.0f. PMID 23168789
- [Background] Andreoli L, Chighizola CB, Banzato A, Pons-Estel GJ, Ramire de Jesus G, Erkan D. Estimated frequency of antiphospholipid antibodies in patients with pregnancy morbidity, stroke, myocardial infarction, and deep vein thrombosis: a critical review of the literature. Arthritis Care Res (Hoboken). 2013 Nov;65(11):1869-73. doi: 10.1002/acr.22066. PMID 23861221
- [Background] Ruiz-Irastorza G, Crowther M, Branch W, Khamashta MA. Antiphospholipid syndrome. Lancet. 2010 Oct 30;376(9751):1498-509. doi: 10.1016/S0140-6736(10)60709-X. Epub 2010 Sep 6. PMID 20822807
- [Background] de Jesus GR, Agmon-Levin N, Andrade CA, Andreoli L, Chighizola CB, Porter TF, Salmon J, Silver RM, Tincani A, Branch DW. 14th International Congress on Antiphospholipid Antibodies Task Force report on obstetric antiphospholipid syndrome. Autoimmun Rev. 2014 Aug;13(8):795-813. doi: 10.1016/j.autrev.2014.02.003. Epub 2014 Mar 17. PMID 24650941
- [Background] Girardi G, Berman J, Redecha P, Spruce L, Thurman JM, Kraus D, Hollmann TJ, Casali P, Caroll MC, Wetsel RA, Lambris JD, Holers VM, Salmon JE. Complement C5a receptors and neutrophils mediate fetal injury in the antiphospholipid syndrome. J Clin Invest. 2003 Dec;112(11):1644-54. doi: 10.1172/JCI18817. PMID 14660741
- [Background] Shamonki JM, Salmon JE, Hyjek E, Baergen RN. Excessive complement activation is associated with placental injury in patients with antiphospholipid antibodies. Am J Obstet Gynecol. 2007 Feb;196(2):167.e1-5. doi: 10.1016/j.ajog.2006.10.879. PMID 17306667
- [Background] Stone S, Pijnenborg R, Vercruysse L, Poston R, Khamashta MA, Hunt BJ, Poston L. The placental bed in pregnancies complicated by primary antiphospholipid syndrome. Placenta. 2006 Apr-May;27(4-5):457-67. doi: 10.1016/j.placenta.2005.04.006. Epub 2005 Jul 6. PMID 16005063
- [Background] Lockshin MD, Kim M, Laskin CA, Guerra M, Branch DW, Merrill J, Petri M, Porter TF, Sammaritano L, Stephenson MD, Buyon J, Salmon JE. Prediction of adverse pregnancy outcome by the presence of lupus anticoagulant, but not anticardiolipin antibody, in patients with antiphospholipid antibodies. Arthritis Rheum. 2012 Jul;64(7):2311-8. doi: 10.1002/art.34402. PMID 22275304
- [Background] Gilbert WM, Nesbitt TS, Danielsen B. The cost of prematurity: quantification by gestational age and birth weight. Obstet Gynecol. 2003 Sep;102(3):488-92. doi: 10.1016/s0029-7844(03)00617-3. PMID 12962929
- [Background] Gnanendran L, Bajuk B, Oei J, Lui K, Abdel-Latif ME; NICUS Network. Neurodevelopmental outcomes of preterm singletons, twins and higher-order gestations: a population-based cohort study. Arch Dis Child Fetal Neonatal Ed. 2015 Mar;100(2):F106-14. doi: 10.1136/archdischild-2013-305677. Epub 2014 Oct 30. PMID 25359876
- [Background] Pijnenborg R, Vercruysse L, Hanssens M. The uterine spiral arteries in human pregnancy: facts and controversies. Placenta. 2006 Sep-Oct;27(9-10):939-58. doi: 10.1016/j.placenta.2005.12.006. Epub 2006 Feb 20. PMID 16490251
- [Background] Redman CW, Sargent IL. Immunology of pre-eclampsia. Am J Reprod Immunol. 2010 Jun;63(6):534-43. doi: 10.1111/j.1600-0897.2010.00831.x. Epub 2010 Mar 23. PMID 20331588
- [Background] Berman J, Girardi G, Salmon JE. TNF-alpha is a critical effector and a target for therapy in antiphospholipid antibody-induced pregnancy loss. J Immunol. 2005 Jan 1;174(1):485-90. doi: 10.4049/jimmunol.174.1.485. PMID 15611274
- [Background] Redecha P, Tilley R, Tencati M, Salmon JE, Kirchhofer D, Mackman N, Girardi G. Tissue factor: a link between C5a and neutrophil activation in antiphospholipid antibody induced fetal injury. Blood. 2007 Oct 1;110(7):2423-31. doi: 10.1182/blood-2007-01-070631. Epub 2007 May 29. PMID 17536017
- [Background] Qing X, Redecha PB, Burmeister MA, Tomlinson S, D'Agati VD, Davisson RL, Salmon JE. Targeted inhibition of complement activation prevents features of preeclampsia in mice. Kidney Int. 2011 Feb;79(3):331-9. doi: 10.1038/ki.2010.393. Epub 2010 Oct 13. PMID 20944547
- [Background] Maynard SE, Min JY, Merchan J, Lim KH, Li J, Mondal S, Libermann TA, Morgan JP, Sellke FW, Stillman IE, Epstein FH, Sukhatme VP, Karumanchi SA. Excess placental soluble fms-like tyrosine kinase 1 (sFlt1) may contribute to endothelial dysfunction, hypertension, and proteinuria in preeclampsia. J Clin Invest. 2003 Mar;111(5):649-58. doi: 10.1172/JCI17189. PMID 12618519
- [Background] Lubbe WF, Butler WS, Palmer SJ, Liggins GC. Fetal survival after prednisone suppression of maternal lupus-anticoagulant. Lancet. 1983 Jun 18;1(8338):1361-3. doi: 10.1016/s0140-6736(83)92141-4. PMID 6134138
- [Background] Branch DW, Scott JR, Kochenour NK, Hershgold E. Obstetric complications associated with the lupus anticoagulant. N Engl J Med. 1985 Nov 21;313(21):1322-6. doi: 10.1056/NEJM198511213132104. PMID 3932854
- [Background] Cowchock FS, Reece EA, Balaban D, Branch DW, Plouffe L. Repeated fetal losses associated with antiphospholipid antibodies: a collaborative randomized trial comparing prednisone with low-dose heparin treatment. Am J Obstet Gynecol. 1992 May;166(5):1318-23. doi: 10.1016/0002-9378(92)91596-3. PMID 1595785
- [Background] Yelnik CM, Laskin CA, Porter TF, Branch DW, Buyon JP, Guerra MM, Lockshin MD, Petri M, Merrill JT, Sammaritano LR, Kim MY, Salmon JE. Lupus anticoagulant is the main predictor of adverse pregnancy outcomes in aPL-positive patients: validation of PROMISSE study results. Lupus Sci Med. 2016 Jan 12;3(1):e000131. doi: 10.1136/lupus-2015-000131. eCollection 2016. PMID 26835148
- [Background] Clark CA, Laskin CA, Spitzer KA. Anticardiolipin antibodies and recurrent early pregnancy loss: a century of equivocal evidence. Hum Reprod Update. 2012 Sep-Oct;18(5):474-84. doi: 10.1093/humupd/dms020. Epub 2012 Jun 13. PMID 22699010